CLINICAL TRIAL: NCT06220058
Title: Comparison Between the Use of a Prophylactic Polypropylene Mesh and the "Small Bites" Technique in Midline Laparotomy Closure for Emergency Colorectal Surgery for Incisional Hernia Prevention
Brief Title: Comparing Polypropylene Mesh and "Small Bites" Technique in Emergency Colorectal Surgery's Midline Laparotomy Closure. Study for Incisional Hernia Prevention.
Acronym: BITEME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fernandez Zamora (Other)
Responsible Party: Sponsor-Investigator, Fernandez Zamora, Principal Investigator, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Organization: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.227
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Incisional Hernia; Wound Infection
Keywords: colorectal cancer; Hernia Incisional; Wound infection; small bites
MeSH Terms: conditions — Colorectal Neoplasms; Incisional Hernia; Wound Infection

STUDY DESIGN:
Masking Description: Patients meeting the inclusion criteria will be randomized 1:1 using random number generation in SPSS v.21, assigning them to either the Mesh or Bites group. Sealed opaque envelopes will be used just before the surgical intervention within the operating room. The envelope will be opened in the operating room upon initiation of midline laparotomy closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Bites (Experimental): Closure of the midline laparotomy using the "small bites" technique
  Interventions: Procedure: Closure of the midline laparotomy using the "small bites" technique
- Group Mesh (Experimental): Closure of the midline laparotomy using the "small bites" technique adding a suprapubic polypropylene mesh.
  Interventions: Procedure: Closure of the midline laparotomy using the "small bites" technique with an absorbable PP mesh

INTERVENTIONS:
Procedure: Closure of the midline laparotomy using the "small bites" technique — Closure of the midline laparotomy using the "small bites" technique will involve employing a monofilament polydioxanone suture with a gauge of 0 (PDS® II Ethicon, Bridgewater, NJ). No Redon drainage system will be left in the subcutaneous tissue.
  Arms: Group Bites
Procedure: Closure of the midline laparotomy using the "small bites" technique with an absorbable PP mesh — Closure of the midline laparotomy using the "small bites" technique will involve employing a monofilament polydioxanone suture with a gauge of 0 (PDS® II Ethicon, Bridgewater, NJ). A partially absorbable low-density polypropylene suprapubic mesh (Ultrapro®, Ethicon) will be added. Mesh fixation will be done with absorbable staples (Ethicon SecurestrapTM) +/- slow-absorbing resorbable sutures at the discretion of the surgical team.
  In the case of a diverting stoma, the prophylactic mesh will not encircle it. A Redon-type drainage will be left at the subcutaneous tissue level. One or two drains will be left at the discretion of the surgical team. Closure of the subcutaneous tissue will be performed with 2/0 or 3/0 absorbable, multifilament, interlocking sutures.
  Arms: Group Mesh

SUMMARY:
The 2023 World Journal of Emergency Surgery guidelines couldn't provide a recommendation for emergency abdominal wall closure due to insufficient consensus (>80% required). Available evidence, predominantly retrospective and heterogeneous, lacks differentiation between urgent and elective colorectal surgeries. Therefore, we advocate for a study comparing laparotomy closures in emergency colorectal surgery to contribute evidence on incisional hernia incidence and subsequent complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colorectal pathology requiring urgent surgical treatment via midline laparotomy.
* Patients undergoing urgent laparoscopic surgery but necessitating conversion to midline laparotomy.
* Urgent surgical intervention required at the level of the colon and/or rectum, even in the presence of other abdominal pathologies.
* Age over 18 years.
* Signed informed consent (IC) from the patient and the investigator.

Exclusion Criteria:

* Severe chronic obstructive pulmonary disease (COPD) according to the GOLD classification or decompensated COPD.
* BMI ≥ 35 kg/m2.
* Re-laparotomies.
* Patients with psychiatric illnesses, addictions, or any disorder hindering the understanding of the Informed Consent.
* Inability to read or comprehend any of the languages in the Informed Consent (Catalan, Spanish).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of incisional hernia. | One year surgery
  Compare the incidence of midline laparotomy incisional hernia at one year post-surgery between the two groups: midline laparotomy closure using the "small bites" technique vs. midline laparotomy closure using the "small bites" technique supplemented with a suprapubic polypropylene mesh.

SECONDARY OUTCOMES:
Incidence of wound infection | 30 postoperative days
  Compare the surgical wound infection rate at 30 days post-surgery, postoperative complications hindering subsequent treatment, as well as comorbidity related to surgical wound infection and rates of parastomal hernias.
Morbidity and mortality rates | 90 postoperative days
  Compare morbidity and mortality between the two groups: initiation of tolerance to a solid oral diet and initiation of ambulation, anastomotic dehiscence, reinterventions, complications according to the Clavien-Dindo classification at 30 and 90 days, and mortality at 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorectal Surgery Section, Department of General and Digestive Surgery, University Hospital of Girona,, Girona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No